CLINICAL TRIAL: NCT05848492
Title: Efficacy of Prophylactic Fluconazole Therapy in Preterm and Very Low Birth Weight Neonates in Preventing Invasive Fungal Infection.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Principal Investigator, Muhammad Tauseef Omer, Post-graduate resident, Services Institute of Medical Sciences, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FluconazolePreterm1
Record Dates: First submitted 2023-04-27; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-04

CONDITIONS: Invasive Candidiases
MeSH Terms: conditions — Candidiasis, Invasive | interventions — Fluconazole; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Prophylactic Fluconazole (Experimental): 12 mg/Kg loading dose of fluconazole given intravenously followed by 6 mg/Kg every 48 hours till 14 days of life, and then 6 mg/kg/day thereafter, for a total duration of 6 weeks (42 days).
  Interventions: Drug: Fluconazole
- placebo group (Placebo Comparator): Normal Saline 2cc given intravenously
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Fluconazole — Fluconazole will be given for prevention of invasive candidiasis in preterm and very low birthweight babies.
  Arms: Prophylactic Fluconazole
Drug: Saline — 0.9% Saline 2cc intravenous will be given to preterm babies in placebo group.
  Arms: placebo group

SUMMARY:
Invasive fungal infection is detecting candida species in blood, cerebrospinal fluid, or urine. Clinical signs of invasive candidiasis may include lethargy, temperature instability, feeding intolerance, apnea, hypotension, respiratory distress, abdominal distension, and thrombocytopenia. Fungal infection has been associated with an increased risk of retinopathy of prematurity and chronic lung disease. Preterm and low birth weight infants have an immature immune system that predisposes them to infections with bacteria, viruses, and fungi. These infants usually require prolonged admission in the neonatal unit and there is often a need for the administration of broad-spectrum antibiotics which predisposes them to colonization with fungi that may invade to cause systemic disease8. Other risk factors for the development of invasive fungal infection include endotracheal intubation, abdominal surgery, the presence of a central venous catheter, administration of H2 antagonists, and steroids. Infection with Candida species is the third most common cause of bloodstream infection in premature infants. Mortality in preterm infants due to invasive candidiasis is around 20% and can be as high as 50% in infants weighing <1500g at birth. Invasive candidiasis is the second most common infectious cause of death in extremely preterm infants. The present study was conducted to determine the incidence of invasive candidiasis among preterm and very low birth weight infants in our neonatal unit and to evaluate the efficacy of prophylactic fluconazole in preventing invasive fungal infection. Based on the results of the present study institutional guidelines may be designed in our neonatal unit relating to antifungal prophylaxis in preterm and very low birth weight infants.

ELIGIBILITY:
Inclusion Criteria:

* Preterm babies born less than 34 weeks of gestation
* very low birth weight babies (weighing < 1500 g at birth)
* Babies <72 hours of age

Exclusion Criteria:

* Babies >72 hours of life
* Syndromic babies
* Babies with suspected metabolic disorders

Ages: 1 Hour to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Invasive candidiases | 2 weeks
  Positive blood, cerebrospinal fluid, or urine culture for candida species will be regarded as invasive candidiasis.

CONTACTS AND LOCATIONS:
Overall Officials: M Tauseef Omer, MBBS FCPS Pediatrics, Principal Investigator — Services Hospital, Lahore
Locations (1):
- Services Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No